CLINICAL TRIAL: NCT01148017
Title: A Phase IIIb, Open-Label, Controlled, Multi-Center Study to Evaluate the Persistence Of Antibody Responses Among Children Who Previously Received Novartis MenACWY Conjugate Vaccine
Brief Title: Evaluation of Meningococcal Immune Response Among Children Who Previously Received MenACWY Conjugate Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: V59P14E1
Record Dates: First submitted 2010-06-16; First posted 2010-06-22 (Estimated); Results first posted 2014-05-14 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-07

CONDITIONS: Meningococcal Meningitis
Keywords: Meningococcal; ACWY; Conjugate Vaccine; Meningitis; Children; Persistence; Booster dose
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ACWY - 4 (Experimental): Subjects who had previously received 4 doses of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in the parent study during their first year of life are administered one booster dose of the same vaccine at 60 months of age.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- ACWY - 2 (Experimental): Subjects who had previously received 1 or 2 doses of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine in the parent study during their second year of life, are administered one booster dose of the same vaccine at 60 months of age.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- Naïve - 40 (Other): Control subjects, age-matched with the intervention groups subjects (40 months of age), to receive 1 optional dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine
- Naïve - 60 (Active Comparator): Control subjects, age-matched with the intervention groups subjects (60 months of age), are administered one dose of Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine.
  Interventions: Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal (groups A, C, W, and Y) oligosaccharide diphtheria CRM-197 conjugate vaccine

SUMMARY:
The primary objective was to evaluate the persistence of bactericidal antibodies in children 40 and 60 months of age previously enrolled in the V59P14 (NCT00474526) study who received Novartis MenACWY Conjugate Vaccine. The study also enrolled age-matched subjects who have never received any meningococcal vaccine (naïve subjects) to serve as a control group. In addition, the response of a booster dose at 60 months was evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Children eligible to be enrolled in the study are those whose parents provide written informed consent, and are in generally good health based on the clinical judgment of the investigators.
* Group 1 and 2 (Follow up) subjects must be 40 +/- 3 months of age at the time of enrollment and participated in the original V59P14 study (NCT00474526).
* Group 3 and 4 (Naïve) subjects must be healthy, meningococcal vaccine-naïve children ages 40 +/- 3 months (Group 3) or 60 +/-3 months (Group 4) at the time of enrollment, respectively.

Exclusion Criteria:

* Serious, acute, or chronic illnesses are reasons for exclusion.
* Subjects who have received any vaccine (excluding influenza vaccines) 28 days preceding enrollment visit. Influenza vaccines (including FluMist®) are excluded for the 14 days prior to the enrollment visit.
* Subjects who have received any meningococcal vaccine since birth (Groups 3 & 4 -naive) or last study dose in V59P14 (NCT00474526) trial (Groups 1 & 2 - follow on).

Ages: 37 Months to 63 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 433 (Actual)
Dates: Start 2010-07; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines, Study Chair — Novartis Vaccines
Locations (19):
- United States (19):
  - Alabama Clinical Therapeutics 806 St. Vincent's Drive, Suite 615, Birmingham, Alabama
  - Premier Health Research 9317 Firestone Blvd., Downey, California
  - Kaiser Permanente Oakland 3505 Broadway, 6th Floor, Room 624, Oakland, California
  - Center for Clinical Trials, LLC 16415 S. Colorado Ave., Suite 308, Paramount, California
  - Center for Clinical Trials, LLC 16660 Paramount Blvd., Suite 301, Paramount, California
  - Kaiser Permanente Pleasanton 7601 Stoneridge Drive, Second Floor, Pleasanton, California
  - Kaiser Permanente San Francisco 2200 O'Farrell St., Sixth Floor, San Francisco, California
  - Kaiser Permanente Santa Clara 710 Lawrence Expressway, Pediatric Clinic Department, Santa Clara, California
  - Children's Memorial Hospital 2300 Children's Plaza, Box 155, Chicago, Illinois
  - Kentucky Pediatric/Adult Research 201 South Fifth Street, Suite 102, Bardstown, Kentucky
  - 28 Annapolis Pediatrics, 200 Forbes Street, Suite 200, Annapolis, Maryland
  - Senders Pediatrics 2054 South Green Road, Cleveland, Ohio
  - Pediatric Medical Associates 160 West Germantown Pike Suite D2, East Norriton, Pennsylvania
  - Children's Health Care 2501 West 12th Street, Erie, Pennsylvania
  - Pennridge Pediatric Associates 270 Main Street, Harleysville, Pennsylvania
  - Kid's Way Pediatrics 3068 Innovation Way, Hermitage, Pennsylvania
  - Pediatric Medical Associates 1077 Rydal Road Suite 300, Rydal, Pennsylvania
  - Pennridge Pediatric Associates 711 Lawn Avenue, Sellersville, Pennsylvania
  - PEAK Research 2859 Washington Rd., Ste. 412B, Upper Saint Clair, Pennsylvania

REFERENCES:
- [Derived] Klein NP, Block SL, Essink B, Barbi S, Smolenov I, Keshavan P. Antibody persistence and booster response following MenACWY-CRM vaccination in children as assessed by two different assay methods. Vaccine. 2019 Jul 26;37(32):4460-4467. doi: 10.1016/j.vaccine.2019.06.076. Epub 2019 Jul 3. PMID 31279564

RESULTS

PARTICIPANT FLOW:
Groups:
- ACWY - 4: Subjects who had previously received 4 doses of MenACWY-CRM in the parent study during their first year of life, are administered one booster dose of the same vaccine at 60 months of age.
- ACWY - 2: Subjects who had previously received 1 or 2 doses of MenACWY-CRM in the parent study during their second year of life, are administered one booster dose of the same vaccine at 60 months of age.
- Naïve - 40: Control subjects, age-matched with the intervention groups subjects (40 months of age), to receive 1 optional dose of MenACWY-CRM.
- Naïve - 60: Control subjects, age-matched with the intervention groups subjects (60 months of age), are administered one dose of MenACWY-CRM.
Period: Overall Study
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40 | Naïve - 60
Started | 214 | 121 | 53 | 45
Completed | 134 | 87 | 53 | 45
Not Completed | 80 | 34 | 0 | 0
Not completed — Withdrawal by Subject | 31 | 14 | 0 | 0
Not completed — Lost to Follow-up | 23 | 10 | 0 | 0
Not completed — Inappropriate enrollment | 1 | 0 | 0 | 0
Not completed — Administrative reason | 22 | 9 | 0 | 0
Not completed — Unable to classify | 3 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was done on the all enrolled population, ie, all subjects who had signed an informed consent, undergone screening procedures, and were enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40 | Naïve - 60 | Total
Number analyzed (Participants) | 214 | 121 | 53 | 45 | 433
Age, Continuous [Mean (Standard Deviation); unit: Months]
  40 months enrollment (N=210, 119, 53, 382) | 39.2 (1.8) | 39.3 (1.7) | 38.7 (1.8) | NA (NA) — Subjects in this group were enrolled at 60 months of age. | 39.2 (1.8)
  60 months enrollment (N=136, 89, 45, 270) | 59.7 (2.2) | 59.6 (2.4) | NA (NA) — Subjects in this group were enrolled at 40 months of age. | 60 (1.7) | 59.7 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 55 | 29 | 26 | 207
  Male | 117 | 66 | 24 | 19 | 226
Region of Enrollment [Number; unit: participants]
  United States | 214 | 121 | 53 | 45 | 433

OUTCOME MEASURES:

1. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Titers ≥ 1:8 Directed Against N. Meningitidis Serogroups A, C, W-135, and Y
Description: The persistence of the antibody response in subjects of 40 months of age, previously vaccinated with MenACWY-CRM in the parent study, and baseline antibody levels in age-matched naive subjects, is measured by the percentage of subjects with human Serum Bactericidal Assay (hSBA) titers ≥ 1:8 directed against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 9 (continuation from the parent study), 40-month visit.
Population: Analysis was done on the Per Protocol Set 40-month persistence (PPS 40-month persistence), ie, all subjects in the enrolled population who provided an evaluable serum sample at the 40-months of age visit and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40
Number analyzed (Participants) | 206 | 117 | 51
Percentages of subjects
  Men A | 10 [6 to 15] | 35 [26 to 44] | 2 [0.05 to 10]
  Men C (N=206, 116, 51) | 34 [28 to 41] | 51 [41 to 60] | 12 [4 to 24]
  Men W-135 (N=204, 115, 51) | 76 [70 to 82] | 83 [74 to 89] | 47 [33 to 62]
  Men Y (N=205, 116, 51) | 67 [60 to 73] | 71 [62 to 79] | 22 [11 to 35]

2. Primary Outcome: Percentages of Subjects With Human Serum Bactericidal Assay (hSBA) Titers ≥ 1:8 Directed Against N. Meningitidis Serogroups A, C, W-135, and Y
Description: The persistence of the antibody response in subjects of 60 months of age previously vaccinated with MenACWY-CRM in the parent study, and baseline antibody levels in age-matched naive subjects, is measured by the percentages of subjects with human Serum Bactericidal Assay (hSBA) titers ≥ 1:8 directed against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 10, 60 months of age
Population: Analysis was done on the Per Protocol Set 60-Month persistence (PPS 60-Month persistence), ie, all subjects in the enrolled population who provided an evaluable serum sample at the 60-month of age visit and had no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 123 | 80 | 45
Percentages of subjects
  Men A | 6 [2 to 11] | 25 [16 to 36] | 2 [0.056 to 12]
  Men C | 27 [19 to 36] | 43 [32 to 54] | 22 [11 to 37]
  Men W-135 (N=121, 78, 45) | 69 [60 to 77] | 74 [63 to 84] | 40 [26 to 56]
  Men Y (N=122, 80, 44) | 56 [46 to 65] | 69 [57 to 79] | 25 [13 to 40]

3. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 Against N Meningitidis Serogroups A, C, W-135, and Y in Subjects of 40 Months of Age
Description: The persistence of the antibody response in subjects of 40 months of age previously vaccinated with MenACWY-CRM in the parent study, and baseline antibody levels in age-matched naive subjects, is measured by the percentage of subjects with human Serum Bactericidal Assay (hSBA) titers ≥ 1:4 directed against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 9, 40 months of age.
Population: Analysis was done on the PPS 40-month persistence.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40
Number analyzed (Participants) | 206 | 117 | 51
Percentages of subjects
  Men A | 13 [9 to 18] | 40 [31 to 50] | 2 [0.05 to 10]
  Men C (N=206, 116, 51) | 43 [36 to 50] | 61 [52 to 70] | 16 [7 to 29]
  Men W-135 (N=204, 115, 51) | 81 [75 to 86] | 88 [80 to 93] | 49 [35 to 63]
  Men Y (N=205, 116, 51) | 76 [69 to 81] | 80 [72 to 87] | 24 [13 to 37]

4. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:4 Against N Meningitidis Serogroups A, C, W-135, and Y Subjects of 60 Months of Age
Description: The persistence of the antibody response in subjects of 60 months of age previously vaccinated with MenACWY-CRM in the parent study, and baseline antibody levels in age-matched naive subjects, is measured by the percentage of subjects with human Serum Bactericidal Assay (hSBA) titers ≥ 1:4 directed against N. meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 10, 60 months of age.
Population: Analysis was done on the PPS 60-Month persistence.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 123 | 80 | 45
Percentages of subjects
  Men A | 9 [5 to 15] | 33 [22 to 44] | 2 [0.056 to 12]
  Men C | 46 [37 to 55] | 60 [48 to 71] | 33 [20 to 49]
  Men W-135 (N=121, 78, 45) | 74 [66 to 82] | 83 [73 to 91] | 42 [28 to 58]
  Men Y (N=122, 80, 44) | 65 [56 to 73] | 74 [63 to 83] | 25 [13 to 40]

5. Secondary Outcome: hSBA Geometric Mean Titers (GMTs) Directed Against N. Meningitidis Serogroups A, C, W-135, and Y in Subjects of 40 Months of Age
Description: The persistence of the antibody response in children of 40 months of age previously vaccinated with MenACWY-CRM in study V59P14 (NCT00474526), and baseline antibody levels in age-matched naive subjects, is measured by the hSBA GMTs directed against N meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 9 (continuation from the parent study), 40-months of age.
Population: Analysis was done on the PPS 40-month persistence.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40
Number analyzed (Participants) | 206 | 117 | 51
Titers
  Men A | 2.54 [2.23 to 2.9] | 4.81 [4.06 to 5.69] | 2.02 [1.57 to 2.61]
  Men C (N=206, 116, 51) | 6.14 [4.98 to 7.59] | 9.24 [7.05 to 12] | 2.52 [1.68 to 3.78]
  Men W-135 (N=204, 115, 51) | 26 [21 to 32] | 29 [22 to 39] | 8.25 [5.47 to 12]
  Men Y (N=205, 116, 51) | 16 [13 to 20] | 18 [14 to 24] | 3.69 [2.44 to 5.57]

6. Secondary Outcome: hSBA GMTs Directed Against N Meningitidis Serogroups A, C, W-135, and Y in Subjects of 60 Months of Age
Description: The persistence of the antibody response in children of 60 months of age previously vaccinated with MenACWY-CRM in study V59P14 (NCT00474526), and baseline antibody levels in age-matched naive subjects is measured by the hSBA GMTs directed against N meningitidis serogroups A, C, W-135, and Y.
Time Frame: Visit 10, 60 months of age.
Population: Analysis was done on the PPS 60-Month persistence.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 123 | 80 | 45
Titers
  Men A | 2.27 [1.95 to 2.63] | 3.74 [3.12 to 4.48] | 2.14 [1.68 to 2.74]
  Men C | 5.17 [3.96 to 6.75] | 9.26 [6.71 to 13] | 3.87 [2.5 to 5.98]
  Men W-135 (N=121, 78, 45) | 17 [13 to 22] | 20 [14 to 28] | 6.63 [4.25 to 10]
  Men Y (N=122, 80, 44) | 11 [8.1 to 14] | 14 [9.94 to 19] | 4.1 [2.61 to 6.45]

7. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ 1:8, and ≥ 1:4 Directed Against N. Meningitidis Serogroups A, C, W-135, and Y, at 1 Month Post-vaccination
Description: The antibody response to one booster dose of MenACWY-CRM in children of 60 months of age who had previously received at least one dose of MenACWY-CRM in the parent study compared to the antibody response to one dose of MenACWY-CRM in meningococcal vaccine-naïve subjects, is measured by the percentage of subjects with hSBA titers ≥ 1:8 and ≥1:4 directed against N. meningitidis serogroups A, C, W-135, and Y, at 1 month post-vaccination.
Time Frame: Visit 11, 1 month after vaccination.
Population: Analysis was done on the PPS-Immunogenicity after one dose of MenACWY-CRM (PPS Post-MenACWY-CRM), ie, all subjects in the enrolled population who correctly received the vaccine, provided at least one evaluable serum sample at the relevant time points and whose assay result was available for at least one serogroup with no major protocol deviation.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 116 | 76 | 45
Percentages of subjects
  Men A (≥1:8) | 97 [91 to 99] | 97 [91 to 100] | 87 [73 to 95]
  Men C (≥1:8; N=115, 75, 45) | 96 [90 to 99] | 99 [93 to 100] | 84 [71 to 94]
  Men W-135 (≥1:8; N=104, 70, 44) | 100 [97 to 100] | 100 [95 to 100] | 89 [75 to 96]
  Men Y (≥1:8; N=111, 74, 44) | 100 [97 to 100] | 100 [95 to 100] | 73 [57 to 85]
  Men A (≥1:4) | 97 [91 to 99] | 97 [91 to 100] | 89 [76 to 96]
  Men C (≥1:4; N=115, 75, 45) | 97 [93 to 99] | 100 [95 to 100] | 87 [73 to 95]
  Men W-135 (≥1:4; N=104, 70, 44) | 100 [97 to 100] | 100 [95 to 100] | 91 [78 to 97]
  Men Y (≥1:4; N=111, 74, 44) | 100 [97 to 100] | 100 [95 to 100] | 80 [65 to 90]

8. Secondary Outcome: Percentage of Subjects With Seroresponse at 1 Month Post-vaccination
Description: The antibody response to one booster dose of MenACWY-CRM in children of 60 months of age who had previously received at least one dose of MenACWY-CRM in the parent study, compared to the antibody response to one dose of MenACWY-CRM in meningococcal vaccine-naïve subjects, is measured by the percentage of subjects with seroresponse at 1 month post-vaccination.
  Seroresponse is defined as hSBA ≥ 1:8 for subjects with pre-vaccination hSBA titer ≤1:4, and as at least a four-fold rise in hSBA for subjects with pre-vaccination hSBA titer ≥ 1:4.
Time Frame: Visit 11, 1 month after vaccination.
Population: Analysis was done on the PPS Post-MenACWY-CRM.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 116 | 76 | 45
Percentage of subjects
  Men A | 97 [91 to 99] | 96 [89 to 99] | 87 [73 to 95]
  Men C (N=115, 75, 45) | 87 [79 to 93] | 87 [77 to 93] | 73 [58 to 85]
  Men W-135 (N=104, 70, 44) | 99 [95 to 100] | 100 [95 to 100] | 57 [41 to 72]
  Men Y (N=111, 74, 44) | 98 [94 to 100] | 99 [93 to 100] | 52 [37 to 68]

9. Secondary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events (AEs) and Other Indicators of Reactogenicity
Description: Number of subjects reporting solicited local and systemic Adverse Events (AEs) and other indicators of reactogenicity after receiving study vaccination.
  Note: solicited AEs were not recorded for naive subjects at 40 months of age, but only SAEs and medically attended AEs.
Time Frame: From day 1 to 7 after vaccination.
Population: Analysis was done on the Solicited Safety Set (from 6 hours to day 7), ie, all subjects who received a vaccination at 60 months and provided postvaccination solicited safety data.
Measure: Number; unit: Subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 60
Number analyzed (Participants) | 129 | 83 | 49
Subjects
  Any local | 67 | 44 | 29
  Injection site pain | 54 | 33 | 24
  Injection site erythema | 26 | 20 | 13
  Injection site induration | 18 | 14 | 10
  Any systemic | 45 | 26 | 23
  Change in eating habits | 14 | 5 | 4
  Sleepiness | 20 | 9 | 7
  Irritability | 24 | 14 | 8
  Vomiting | 4 | 0 | 3
  Diarrhea | 7 | 1 | 1
  Arthralgia | 2 | 4 | 0
  Headache | 6 | 6 | 2
  Rash | 4 | 2 | 3
  Fever | 4 | 2 | 2
  Any other | 18 | 11 | 7
  Stayed home due to reaction | 5 | 0 | 0
  Use of analgesics/antipyretics | 18 | 11 | 7

10. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs and SAEs
Description: Number of subjects reporting unsolicited AEs, serious adverse events (SAEs) and medically attended AEs after receiving study vaccination.
Time Frame: Day 1 to 7 after vaccination for any unsolicited AEs, day 1 to study termination for SAEs and medically attended AEs (for the naive-40 group), day 8 to study termination for SAEs and medically attended AEs (for the other groups).
Population: Analysis was done on the Post MenACWY at 60 months safety set ie, all subjects who received a vaccination at 60 months and were assessed for postvaccination safety, and on the Post MenACWY at 40 Months Safety Set, ie, the Naive subjects enrolled at 40 months of age who received vaccination at 40 months and were assessed for post vaccination safety.
Measure: Number; unit: Number of subjects
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40 | Naïve - 60
Number analyzed (Participants) | 132 | 87 | 11 | 50
Number of subjects
  Any unsolicited AE | 7 | 8 | NA — Unsolicited AEs were not recorded for this group. | 12
  Medically attended AEs | 0 | 0 | 27 | 0
  Any SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs were collected from day 1 to day 7 after vaccination. Serious AEs were collected from day 1 to study termination for the naive-40 group, and from day 8 to study termination for the other groups.
Description: Analysis for the solicited and unsolicited non-serious AEs was done on the Overall Post MenACWY Safety Set, ie, all subjects who received a vaccination at 40 or 60 months and were assessed for postvaccination safety. Analysis for serious adverse events was done on the Post MenACWY at 60 Months and at 40 Months Safety Sets.
Arm/Group | ACWY - 4 | ACWY - 2 | Naïve - 40 | Naïve - 60
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/87 | 0/11 | 0/50
Other Adverse Events (participants affected / at risk) | 86/132 | 57/87 | 3/11 | 39/50
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ACWY - 4 (N=132) | ACWY - 2 (N=87) | Naïve - 40 (N=11) | Naïve - 60 (N=50)
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 2 | 0 | 1
Vomiting (Gastrointestinal disorders) | 4 | 0 | 0 | 3
Injection site erythema (General disorders) | 26 | 22 | 0 | 13
Injection site induration (General disorders) | 21 | 15 | 0 | 11
Injection site pain (General disorders) | 59 | 37 | 0 | 24
Irritability (General disorders) | 24 | 14 | 0 | 9
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 2
Viral pharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 1 | 1
Headache (Nervous system disorders) | 6 | 7 | 0 | 2
Somnolence (Nervous system disorders) | 21 | 9 | 0 | 7
Eating disorders (Psychiatric disorders) | 14 | 5 | 0 | 4
Ingrown nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 4 | 2 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No